CLINICAL TRIAL: NCT02650284
Title: A Prospective, Randomised Controlled Trial Evaluating Total Knee Replacement With the Stryker Triathlon Primary Total Knee System Performed Using Stryker's Robotic-arm Assisted Surgery System, Mako, Compared to Bicompartmental Knee Replacement With Restoris MCK Multicompartmental Knee System Performed Using Stryker's Robotic-arm Assisted Surgery System, Mako
Brief Title: A Trial Evaluating TKR Compared to BKR Performed Using Stryker's Mako Robot
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Participant recruitment difficulties. Ruling to terminate study made Oct 2019
Sponsor: Stryker South Pacific (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAKORCT-15
Record Dates: First submitted 2016-01-06; First posted 2016-01-08 (Estimated); Results first posted 2021-06-04 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Non-inflammatory Degenerative Joint Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bicompartmental Knee Replacement (BKR) (Other): Receiving Restoris MCK Multicompartmental Knee System for Bicompartmental Knee Replacement (BKR). Surgery performed using Stryker's robotic-arm assisted surgery system Mako
  Interventions: Device: Restoris MCK Multicompartmental Knee System
- Total Knee Replacement (TKR) (Other): Receiving Stryker Triathlon Primary Total Knee System for Total Knee Replacement. Surgery performed using Stryker's robotic-arm assisted surgery system Mako
  Interventions: Device: Stryker Triathlon Primary Total Knee System

INTERVENTIONS:
Device: Stryker Triathlon Primary Total Knee System — Total Knee Replacement
  Arms: Total Knee Replacement (TKR)
Device: Restoris MCK Multicompartmental Knee System — Bicompartmental Knee Replacement
  Arms: Bicompartmental Knee Replacement (BKR)

SUMMARY:
A prospective, randomised controlled trial evaluating Total Knee Replacement with the Stryker Triathlon Primary Total Knee System, compared to Bicompartmental Knee Replacement with Restoris MCK Multicompartmental Knee System performed using Stryker's Robotic-arm assisted surgery system, Mako.

DETAILED DESCRIPTION:
This study is a prospective, randomised clinical study comparing clinical outcomes of Knee Replacement using the Oxford Knee Score (OKS), in patients receiving either Bicompartmental Knee Replacement performed using Stryker's robotic-arm assisted surgery system Mako, to Total Knee Replacement using the Triathlon Total Knee System performed with either conventional instrumentation or navigation. Functional and radiographic outcomes will be additionally collected as part of this study.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is a suitable candidate for a Bicompartmental Knee Replacement and has moderate to severe patellofemoral wear and medial compartment wear (surgeons discretion)
2. The patient has no fixed flexion greater than 10 degrees.
3. The patient has maximal flexion greater than 100 degrees
4. The patient has a passively correctable varus deformity
5. The patient has a functionally Intact Anterior Cruciate Ligament (ACL.)
6. The patient has no significant patellofemoral malalignment
7. The patient has negligible lateral compartment degeneration with no appreciable loss of cartilage height (surgeon's discretion).
8. The patient has pain that is not localised to the medial compartment only
9. The patient is a male or non-pregnant female.
10. The patient has signed the study specific, Human Research Ethics Committee (HREC)- approved Informed Consent document and is willing and able to comply with the specified pre-operative and post-operative clinical and radiographic evaluations

Exclusion Criteria:

1. The patient has a clinically deficient ACL and cruciate and collateral ligament insufficiency on CT arthrogram.
2. The patient is undergoing revision surgery
3. The patient has greater than 10° of hyperextension, greater than 10° of varus or valgus deformity, greater than 10° Flexion Contracture
4. The patient has active, local infection or previous intra-articular infection
5. The patient has skeletal immaturity
6. The patient is without sufficient bone stock to allow appropriate insertion and fixation of the prosthesis
7. The patient's weight, age or activity level might cause extreme loads and early failure of the system (surgeons discretion).
8. The patient has a systemic or local condition that would limit the ability to assess the performance of the device e.g. neuromuscular or neurosensory deficiency, disorder leading to progressive bone deterioration (including rheumatoid arthritis and osteoporosis), or patient is immunologically suppressed.
9. Patient has a cognitive impairment, an intellectual disability or a mental illness that is considered by the investigator to inhibit the patient's capacity to consent to research and the ability to participate in it
10. Patients with tricompartmental disease are contraindicated from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-08-12 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Clark, Dr, Principal Investigator — Perth Hip and Knee and St John of God Hospital
Locations (1):
- Perth Hip & Knee, Subiaco, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Upon being assessed against the inclusion and exclusion criteria, suitable patients were randomised to one arm of the study.
Pre-assignment Details: In addition to the 8 Bicompartmental and 9 Total Knee replacement patients, 1 patient in the study was not randomised prior to surgery.
Period: Overall Study
Arm/Group | Bicompartmental Knee Replacement (BKR) | Total Knee Replacement (TKR)
Started | 8 | 9
Completed | 5 | 5
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 3 | 3
Not completed — Consent incorrectly taken | 0 | 1

BASELINE CHARACTERISTICS:
Population: 1 patient in the Total Knee study arm was consented incorrectly and their data could not be used in analyses (i.e. reducing the number of participants in this study arm to 8).
Groups:
- Total: Total of all reporting groups
Arm/Group | Bicompartmental Knee Replacement (BKR) | Total Knee Replacement (TKR) | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (4.56) | 64.0 (4.85) | 65 (4.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 5 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Oxford Knee Score
Description: Comparing clinical outcomes using the Oxford Knee Score. The OKS is a participant completed 12 question form on activities of daily living that assess function and pain. Scores can range from 0 to 48 with lower scores indicating a poor outcome and higher scores indicating a more satisfactory joint outcome.
Time Frame: pre-op, 6 weeks, 3 months, 12 months, 24 months
Population: The number of recruited patients did not reach the required sample size. 1 patient in the Total Knee study arm was consented incorrectly and their data could not be used in analyses (i.e. reducing the number of participants in this study arm to 8).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bicompartmental Knee Replacement (BKR) | Total Knee Replacement (TKR)
Number analyzed (Participants) | 8 | 8
units on a scale
  Oxford pre-operative | 22.63 (8.14) | 26.75 (8.90)
  Oxford 6-weeks: number analyzed (Participants) | 8 | 7
  Oxford 6-weeks | 34.00 (6.69) | 30.14 (3.80)
  Oxford 3-months: number analyzed (Participants) | 8 | 7
  Oxford 3-months | 39.00 (3.61) | 33.29 (7.63)
  Oxford 12-months: number analyzed (Participants) | 7 | 6
  Oxford 12-months | 40.43 (4.17) | 40.33 (7.95)
  Oxford 24-months: number analyzed (Participants) | 5 | 4
  Oxford 24-months | 41.20 (5.49) | 43.75 (3.34)
Statistical Analysis 1: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); Comparison between groups at pre-operation timepoint; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.46, t-test, 2 sided — The number of recruited patients did not reach the required sample size. Power score assessments no longer hold, thus there is low confidence in the findings
Statistical Analysis 2: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); Comparison between groups at 6-week timepoint; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.23, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); Comparison between groups at 3-month timepoint; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.10, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); Comparison between groups at 12-month timepoint; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.98, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); Comparison between groups at 24-month timepoint; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.50, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Health Related Quality of Life EQ-5D
Description: Comparing functional and clinical outcomes using the EQ-5D. The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. The participant is asked to indicate his/her health state by indicating the most appropriate level for each of the 5 dimensions. Responses may be converted into a single summary index by applying a formula that essentially attaches values (also called weights) to each of the levels in each dimension. Index values range from 0-1, with 1 being representing "full health". The EQ VAS records the participant's self-rated health on a vertical, visual analogue scale where the endpoints are labelled from 100 ='Best imaginable health state' to 0= 'Worst imaginable health state'. The VAS scales represents health on the day.
Time Frame: 24 months/ 2years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bicompartmental Knee Replacement (BKR) | Total Knee Replacement (TKR)
Number analyzed (Participants) | 8 | 8
units on a scale
  Pre-op EQ-5D Index | 0.16 (0.45) | 0.28 (0.40)
  Pre-op EQ-5D VAS | 78.50 (12.22) | 81.50 (12.21)
  3-month EQ-5D Index: number analyzed (Participants) | 8 | 7
  3-month EQ-5D Index | 0.69 (0.35) | 0.66 (0.31)
  3-month EQ-5D VAS: number analyzed (Participants) | 8 | 7
  3-month EQ-5D VAS | 82.25 (12.67) | 90.00 (13.35)
  12-month EQ-5D Index: number analyzed (Participants) | 6 | 5
  12-month EQ-5D Index | 0.48 (0.41) | 0.65 (0.45)
  12-month EQ-5D VAS: number analyzed (Participants) | 6 | 5
  12-month EQ-5D VAS | 74.50 (10.13) | 89.20 (10.23)
  24-month EQ-5D Index: number analyzed (Participants) | 5 | 4
  24-month EQ-5D Index | 0.63 (0.62) | 0.89 (0.13)
  24-month EQ-5D VAS: number analyzed (Participants) | 5 | 4
  24-month EQ-5D VAS | 80.40 (11.36) | 87.25 (10.62)
Statistical Analysis 1: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare EQ-5D Index preoperatively between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.59, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare EQ-5D index at 3-months between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.90, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare EQ-5D index at 12-months between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.57, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare EQ-5D index at 24-months between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.49, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare EQ-5D VAS preoperatively between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.65, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare EQ-5D VAS at 3-months between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.30, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare EQ-5D VAS at 12-months between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.06, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare EQ-5D VAS at 24-months between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.44, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: VAS Pain
Description: Comparing functional and clinical outcomes using the VAS pain. Pain at rest and pain during mobilization are measured using a 10 centimeter Visual Analogue Scale (VAS). Participants are asked to indicate their level of pain with 0 being no pain and 100 being the worst pain.
Time Frame: 24 months/ 2years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bicompartmental Knee Replacement (BKR) | Total Knee Replacement (TKR)
Number analyzed (Participants) | 8 | 8
units on a scale
  Pre-op VAS Pain at rest: number analyzed (Participants) | 8 | 7
  Pre-op VAS Pain at rest | 36.63 (26.89) | 36.14 (21.91)
  Pre-op VAS Pain at mobilization: number analyzed (Participants) | 8 | 7
  Pre-op VAS Pain at mobilization | 65.00 (25.63) | 56.86 (25.18)
  3-month VAS Pain at rest: number analyzed (Participants) | 6 | 4
  3-month VAS Pain at rest | 12.00 (17.45) | 22.25 (18.46)
  3-month VAS Pain at mobilization: number analyzed (Participants) | 6 | 4
  3-month VAS Pain at mobilization | 23.67 (29.44) | 24.25 (16.41)
  12-month VAS Pain at rest: number analyzed (Participants) | 5 | 4
  12-month VAS Pain at rest | 10.40 (9.41) | 19.00 (32.91)
  12-month VAS Pain at mobilization: number analyzed (Participants) | 5 | 4
  12-month VAS Pain at mobilization | 13.60 (9.65) | 24.25 (34.40)
  24-month VAS Pain at rest: number analyzed (Participants) | 3 | 4
  24-month VAS Pain at rest | 0.67 (0.47) | 3.50 (2.69)
  24-month VAS Pain at mobilization: number analyzed (Participants) | 3 | 4
  24-month VAS Pain at mobilization | 2.33 (1.70) | 7.75 (4.60)
Statistical Analysis 1: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare VAS Pain at Rest preoperatively between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.97, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare VAS Pain at Rest at 3-months between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.45, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare VAS Pain at Rest at 12-months between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.64, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare VAS Pain at Rest at 24-months between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.19, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare VAS Pain at Mobilisation preoperatively between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.57, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare VAS Pain at Mobilisation at 3-months between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.98, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare VAS Pain at Mobilisation at 12-months between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.58, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare VAS Pain at Mobilisation at 24-months between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.16, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: New Knee Society Score (KSS)
Description: Comparing functional and clinical outcomes using the KSS. The Knee Society Clinical Rating System is comprised of two distinct sub-scores: one for pain, range of motion (ROM) and joint stability, and one for functional parameters. Sub-scores range from a minimum score of 0 to a maximum of 100 points. Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome.
Time Frame: 24 months/ 2years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bicompartmental Knee Replacement (BKR) | Total Knee Replacement (TKR)
Number analyzed (Participants) | 8 | 8
units on a scale
  KSS function at pre-operation: number analyzed (Participants) | 7 | 8
  KSS function at pre-operation | 44.29 (9.65) | 48.00 (15.59)
  KSS function at 3-month: number analyzed (Participants) | 8 | 7
  KSS function at 3-month | 76.44 (12.08) | 61.00 (15.34)
  KSS function at 24-month: number analyzed (Participants) | 4 | 3
  KSS function at 24-month | 84.50 (9.39) | 85.33 (10.40)
Statistical Analysis 1: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare New Knee Society Function Score preoperatively between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.62, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare New Knee Society Function Score at 3-months between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.06, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare New Knee Society Function Score at 24-months between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.93, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Forgotten Joint Score (FJS)
Description: Comparing functional and clinical outcomes using the FJS. The Forgotten Joint Score (FJS) is a 12 question form that asks the patient their level of awareness of their artificial joint in 12 scenarios commonly encountered in daily life. Scores can range from 0 to 100 with a higher score indicating a better outcome (high degree of forgetting the joint in everyday life).
Time Frame: 24 months/ 2years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bicompartmental Knee Replacement (BKR) | Total Knee Replacement (TKR)
Number analyzed (Participants) | 8 | 8
units on a scale
  FJS pre-operative: number analyzed (Participants) | 4 | 5
  FJS pre-operative | 11.60 (3.56) | 13.75 (5.53)
  FJS 3-month: number analyzed (Participants) | 8 | 7
  FJS 3-month | 51.30 (25.92) | 30.36 (25.41)
  FJS 12-month: number analyzed (Participants) | 7 | 6
  FJS 12-month | 58.63 (27.04) | 63.19 (32.40)
  FJS 24-month: number analyzed (Participants) | 5 | 4
  FJS 24-month | 64.58 (23.46) | 66.67 (19.60)
Statistical Analysis 1: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); Comparison between groups at pre-operation timepoint; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.57, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare FJS at 3-months between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.17, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare FJS at 12-months between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.80, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare FJS at 24-months between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.90, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

6. Secondary Outcome: Incidence of Loosening, Reoperation and Revision
Description: To compare incidence of loosening, reoperation and revision rates. The incidence (ie number of participants who experienced lossening, reoperation or revision) will be counted and presented as a whole number or percentage of the total number of patients, however they will be identified from analysing Xrays and checking Serious Adverse Event/ Adverse Event reports.
Time Frame: 6 weeks, 3 months, 12 months, 24 months
Population: Image quality not obtained to perform incidence calculations thus the incidence of loosening, reoperation and revision detailed below are solely based off the Serious Adverse Events and Adverse Events reported. 1 patient in the Total Knee study arm was consented incorrectly and their data could not be used in analyses (i.e. reducing the number of participants in this study arm to 8).
Measure: Count of Participants; unit: Participants
Arm/Group | Bicompartmental Knee Replacement (BKR) | Total Knee Replacement (TKR)
Number analyzed (Participants) | 8 | 8
Participants
  Incidence of loosening | 0 | 0
  Incidence of reoperation | 0 | 0
  Incidence of revision | 0 | 0

7. Secondary Outcome: Length of Hospital Stay
Description: To compare length of hospital stay between the two arms of the study
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of nights
Arm/Group | Bicompartmental Knee Replacement (BKR) | Total Knee Replacement (TKR)
Number analyzed (Participants) | 8 | 8
Number of nights | 3 (1.32) | 2.86 (0.64)
Statistical Analysis 1: Comparison: Bicompartmental Knee Replacement (BKR) vs Total Knee Replacement (TKR); To compare length of hospital stay (number of nights) between both groups; Test type: Equivalence — Equivalence defined as less than or equal to 1 standard deviation between the two means; p = 0.81, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 2 years post-operation
Description: 1 patient in the Total Knee study arm was consented incorrectly and their data could not be used in analyses (i.e. reducing the number of participants in this study arm to 8).
Arm/Group | Bicompartmental Knee Replacement (BKR) | Total Knee Replacement (TKR)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 3/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bicompartmental Knee Replacement (BKR) (N=8) | Total Knee Replacement (TKR) (N=8)
Contralateral knee osteoarthirits (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Contralateral knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Contralateral Bicompartmental Knee Replacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Internal Cardiac Defibrillator implanted (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bicompartmental Knee Replacement (BKR) (N=8) | Total Knee Replacement (TKR) (N=8)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — (operative side)
Lateral knee pain and anterior fat pad impingement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — (operative side)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — (operative side)
Sinus and ear infection (Ear and labyrinth disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
There existed complexities in recruiting patients that complied with the inclusion and exclusion criteria of the study. The randomised nature of this study required detailed criteria, yet it was difficult in recruiting patients suitable for both bicompartmental and total knee replacement surgeries.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Since the study has been discontinued due to the sample size not being reached, the data cannot be analysed and there are no trial results to discuss/ publish.

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT02650284/Prot_SAP_000.pdf
  • Informed Consent Form: Patients receiving CT but NO Arthrogram (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT02650284/ICF_001.pdf
  • Informed Consent Form: Patients receiving CT WITH Arthrogram (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT02650284/ICF_002.pdf